CLINICAL TRIAL: NCT04750161
Title: The Role Of Neutrophil Proteases As Global Regulators Of Il-1 Family Cytokine Activity In Skin Disorders
Acronym: NEUTROPRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Collaborators: Science Foundation Ireland (Other); University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Matthew Coalter, Study Investigator, St. James's Hospital, Ireland
Other Study IDs: CRFSJ0133
Record Dates: First submitted 2021-02-06; First posted 2021-02-11 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Psoriasis Vulgaris; Atopic Dermatitis; Ichthyosis Vulgaris
MeSH Terms: conditions — Dermatitis, Atopic; Ichthyosis Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Psoriasis Vulgaris
  Interventions: Other: No intervention
- Atopic Dermatitis
  Interventions: Other: No intervention
- Ichthyosis Vulgaris
  Interventions: Other: No intervention
- Healthy Controls
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be given to participants. It is purely observational.

SUMMARY:
Pro-inflammatory cytokines are critically important drivers of inflammatory and autoimmune diseases and cytokine-targeted biologics have been transformative in the treatment of several inflammatory and autoimmune diseases. As the diversity of approved cytokine-targeted biologic therapies grows, it will become increasingly important to stratify patients on the basis of specific genetic or disease biomarker phenotypes to ensure that patients receive the appropriate cytokine-targeted biologic, at the appropriate dose, and at the appropriate time. This project aims to explore patterns of pro-inflammatory cytokine/chemokine expression within normal versus (i) psoriatic, (ii) eczematic, (iii) ichthyotic human skin, as well as in human and mouse models of skin inflammation, with the objective of identifying cytokine response profiles ('cytokine fingerprints') that will provide a molecular basis for (a) the stratification of patients into disease subtypes that (b) enable cytokine-directed biologics to be targeted towards patients that are most likely to benefit from them. The investigators anticipate that 'cytokine fingerprinting' will aid in the selection of the most appropriate biologics in patients that are most likely to benefit from such therapies.

DETAILED DESCRIPTION:
Neutrophils, the 'first responder' cells of the immune system are recruited rapidly to sites of infection or inflammation. Neutrophil granule proteases, cathepsin G, elastase and proteinase-3, are thought to function as anti-microbial effectors, cooperatively working to kill microorganisms during infection. However, evidence also suggests that these enzymes play an important role in the coordination and escalation of inflammatory reactions, but how this is achieved has remained obscure. IL-1 family cytokines are important initiators of inflammation but require processing by enzymes for activation. The IL-1 cytokine family is made up of 11 members, but this study will focus on the processing and activation of 7 of these pro-inflammatory cytokines (IL-1a, IL-1b, IL-18, IL-33, IL-36a, IL-36b and IL-36g). Members of the extended IL-1 family are found at high levels in barrier surfaces such as the skin, and thought to play a role in conditions such as psoriasis, atopic dermatitis/eczema and ichthyosis. Psoriasis particularly is associated with massive neutrophil influx. This study aims to investigate the physiological relevance of neutrophil proteases in the activation of IL-1 family cytokines in skin disorders.

The investigators plan to study the contribution of neutrophil proteases to inflammation in normal skin versus lesions from areas of skin affected by the conditions described above. The investigators are interested in measuring the levels of active neutrophil proteases in normal healthy skin versus skin lesions from affected sites compared to non-lesional, unaffected skin. The investigators also are interested to see if levels of neutrophil proteases found in lesions from affected skin sites are able to process and activate IL-1 family cytokines and contribute to inflammation in this way.

The investigators plan to include up to 80 participants; 20 healthy volunteers, 20 participants who will have a diagnosis of psoriasis, 20 participants who have a diagnosis of atopic dermatitis and 20 patients who have a diagnosis of ichthyosis with active lesions on their arms. Skin samples from normal versus lesional and non-lesional, unaffected skin will be taken by tape stripping method.

ELIGIBILITY:
Inclusion Criteria:

* Have psoriasis, atopic Dermatitis or ichthyosis vulgaris with visible skin lesions, preferably on the forearm which are amenable to sampling.
* Healthy control group without any skin disease.

Exclusion Criteria:

* Under 18 years old
* Fully treated skin disease without active lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A mix of participants from all ages and genders, 20 from each inflammatory skin disorders: psoriasis, atopic dermatitis and ichthyosis vulgaris as well as 20 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-03-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Cytokine Profiles | 6 months
  The generation of a large dataset of cytokine profiles from uninvolved versus involved areas of skin from approximately 80 patients displaying heterogenous clinical symptoms.

SECONDARY OUTCOMES:
Develop sampling techniques | 6 months
  To develop practical and minimally invasive ways of generating 'cytokine fingerprints' using tape-stripped skin samples from psoriasis patients, with the ultimate goal of developing such tests into companion diagnostics.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Irvine, Principal Investigator — St. James Hospital
Locations (1):
- Clinical Research Facility, St James Hospital, Dublin, Ireland